CLINICAL TRIAL: NCT06509087
Title: The Combined Utility of Angio-CT and MRI in Managing Chronic Musculoskeletal Pain: a Prospective Study to Evaluate the Efficacy of Transarterial Microembolization
Status: Recruiting | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, yi-chih HSU, Attending doctor, Tri-Service General Hospital
Other Study IDs: C202405040
Record Dates: First submitted 2024-07-08; First posted 2024-07-19 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Chronic Musculoskeletal Disease; Transarterial Embolization; Magnetic Resonance Imaging; Angiography; Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAME responder: Transarterial microembolization (TAME) is performed on all included patients with chronic shoulder or knee joint pain. Responders are determined if pain score reduction is two points or more based on the Visual Analogue Scale (VAS) at 1-month follow-up after the TAME.
  Interventions: Procedure: Transarterial microembolization (TAME)
- TAME non-responder: Transarterial microembolization (TAME) is performed on all included patients with chronic shoulder or knee joint pain. Non-responders are determined if pain score reduction is less than two points or if pain score increases based on the Visual Analogue Scale (VAS) at 1-month follow-up after the TAME.
  Interventions: Procedure: Transarterial microembolization (TAME)

INTERVENTIONS:
Procedure: Transarterial microembolization (TAME) — TAME primarily targets abnormal neovascularization for embolization in chronic shoulder or knee joint pain.

SUMMARY:
Transarterial microembolization (TAME) is a novel treatment option for chronic musculoskeletal pain, especially suitable for patients who have not responded to conservative treatment or are unsuitable for surgical procedures. This minimally invasive technique primarily targets abnormal neovascularization for embolization, relying heavily on precise information provided by various imaging techniques to ensure the effectiveness and safety of the treatment. This study aims to explore the application of integrating preoperative magnetic resonance imaging (MRI) evidence of patient pain and intraoperative high-resolution synchronous imaging information from fused computed tomography (CT) and angiography systems. This integration is intended to enhance preoperative planning, intraoperative guidance, and final treatment outcome assessment, focusing on its crucial contribution to treatment success. It is hoped that this approach will provide pain intervention physicians with reliable diagnostic tools and safe treatment methods, thereby improving treatment outcomes for patients with chronic musculoskeletal pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic musculoskeletal shoulder or knee joint pain in our hospital, including degenerative knee arthritis, adhesive capsulitis of the shoulder, and those confirmed by physical examination or ultrasound-guided injection to have tendinopathy or ligamentopathy, who have failed drug therapy, rehabilitation, or injection treatments, with a duration of symptoms greater than three months, are the target population of this study.

Exclusion Criteria:

* Pregnancy, coagulation disorders, symptoms of relevant local infections or tumors, and patients allergic to contrast agents. Patients must have complete medical records; those who do not meet the inclusion criteria will be excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic musculoskeletal shoulder or knee joint pain who undergo preoperative magnetic resonance imaging (MRI) and receive transarterial microembolization (TAME) performed using fused computed tomography (CT) and angiography systems.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain relief | day 0, day 1, week 1, month 1, month 3, and month 6.
  Pain relief is measured according to the Visual Analog Scale (VAS) immediately prior to (baseline) and after the TAME procedure (day 0) as well as day 1, week 1, month 1, month 3, and month 6.

SECONDARY OUTCOMES:
Functional improvement (for shoulder joint) | day 0, day 1, week 1, month 1, month 3, and month 6.
  Functional improvement is measured according to Shoulder Pain and Disability Index (SPADI) for patients with chronic shoulder pain immediately prior (baseline) to and after the TAME procedure (day 0) as well as day 1, week 1, month 1, month 3, and month 6.
Functional improvement (for knee joint) | day 0, day 1, week 1, month 1, month 3, and month 6.
  Functional improvement is measured according to the Western Ontario and McMaster Universities Arthritis Index (WOMAC) for patients with chronic knee pain immediately prior (baseline) to and after the TAME procedure (day 0) as well as day 1, week 1, month 1, month 3, and month 6.

OTHER OUTCOMES:
The technical success rate of TAME procedure | Immediately after the TAME procedure
  The technical success rate is judged according to the digital subtraction angiography (DSA). A successful procedure is determined by decreased neovascularization via targeted vessels embolization by the fused CT and angiography system.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chih Hsu, M.D., Principal Investigator — Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No